CLINICAL TRIAL: NCT02374086
Title: A Pilot Study to Test the Benefits of Exercise Training in Women With Ischemic Syndrome
Brief Title: Benefits of Exercise Training in Women With Ischemic Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment slower than usual.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO37771
Record Dates: First submitted 2015-02-18; First posted 2015-02-27 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Microvascular Coronary Dysfunction
MeSH Terms: interventions — Exercise

ARMS (1):
- Exercise Training (Experimental): Subjects will exercise for 8 weeks
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training

SUMMARY:
Angina in the absence of obstructive coronary artery disease is highly prevalent in women, and leads to increased risk for major cardiovascular events, including myocardial infarction, stroke, and heart failure. Annual mortality rates are ten-fold higher than mortality from breast cancer, and the lifetime cost of health care for women with non-obstructive chest pain is close to $1 million. Coronary microvascular dysfunction is a major etiological feature of this disease, and may contribute to disease progression. Despite our general understanding, effective treatment remains elusive. This pilot study will test whether regular exercise training can improve/reverse coronary microvascular dysfunction in women with angina but no obstructive coronary artery disease.

DETAILED DESCRIPTION:
We will study 10 women with signs and symptoms of ischemia but no evidence of obstructive coronary artery disease.

Procedures:

Aerobic fitness: Incremental exercise test to volitional exhaustion on a exercise bike to assess the maximal rate of oxygen consumption.

Cardiac magnetic resonance imaging: To assess cardiac morphology and function. Cardiac perfusion imaging: Using MRI, we will assess the rate of uptake of a contrast media (gadolinium) at rest and in response to a vasodilating substance (adenosine) to evaluate myocardial perfusion reserve.

Protocol:

Participants will undergo aerobic fitness testing, cardiac MRI and perfusion imaging at baseline and following 8-weeks of regular exercise training.

ELIGIBILITY:
Inclusion Criteria:

1. Women with persistent chest pain but no obstructive disease (defined as 50% luminal diameter stenosis in >1 epicardial coronary arteries)
2. Fully understanding and willing to undergo study procedures
3. Understanding and willing to sign consent form.

Exclusion Criteria:

1. Acute coronary syndrome (defined by WHO), cardiogenic shock or requiring inotropic or intra-aortic balloon support;
2. Planned percutaneous coronary intervention or coronary artery bypass graft or established obstructive CAD with ischemia eligible for revascularization,
3. Acute myocardial infarction;
4. Patients with concurrent cardiogenic shock or requiring inotropic or intra-aortic balloon support;
5. Prior non-cardiac illness with an estimated life expectancy <4 years;
6. Unable to give informed consent;
7. Allergy or contra-indication to cardiac magnetic resonance imaging, including renal failure, claustrophobia, and asthma, uncontrolled moderate hypertension (sitting blood pressure >160/95 mmHg with measurements recorded on at least 2 occasions), conditions likely to influence outcomes: Severe lung, creatinine >1.8 or CrCl ≤ 50ml/min) or hepatic disease;
8. Contraindications to adenosine or regadensoson (Lexiscan)
9. Surgically uncorrected significant congenital or valvular heart disease and other disease likely to be fatal or require frequent hospitalization within the next six months;
10. Adherence or retention issues;
11. Unwilling to complete follow-up evaluation;
12. Aortic stenosis (valve area <1.5cm);
13. Left ventricular systolic dysfunction (ejection fraction <35%);
14. Taking potent CYP3A4 inhibitors (ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir);
15. Women who are pregnant.
16. Allergy to animal dander.
17. Unable to perform exercise

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in the maximal rate of myocardial oxygen consumption | Change from baseline at 8 weeks

SECONDARY OUTCOMES:
Change in myocardial perfusion reserve index | change from baseline at 8 weeks
Change in left ventricular diastolic function | change from baseline at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes